CLINICAL TRIAL: NCT02911883
Title: Evaluation of the Repeatability and Reproducibility of AngioVue
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-51133
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Normal, Glaucoma & Retinal Pathology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal: Not having glaucoma or retinal pathology
  Interventions: Device: Optical Coherence Tomography Angiography
- Glaucoma: Having glaucoma.
  Interventions: Device: Optical Coherence Tomography Angiography
- Retina: Having retinal pathology
  Interventions: Device: Optical Coherence Tomography Angiography

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography

SUMMARY:
The purpose of this study is to assess the repeatability and reproducibility of measurements of the vascular structures and the anatomical structures of the posterior pole of the eye based on AngioVue volume scans in normal subjects, glaucoma patients, and retina patients.

ELIGIBILITY:
Inclusion Criteria:

1. Normal

   * Age > 18.
   * No retinal pathology or glaucoma.
2. Glaucoma patient

   * Age > 18.
   * Have glaucoma.
3. Retina patient

   * Age > 18.
   * Have retina pathology.

Exclusion Criteria:

1. Normal

   * Unable to complete required exams.
   * Poor quality image data.
2. Glaucoma patient

   * Unable to complete required exams.
   * Poor quality image data.
   * Retinal pathology.
3. Retina patient

   * Unable to complete required exams.
   * Poor quality image data.
   * Glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine or follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Retina vasculature | Day 1